CLINICAL TRIAL: NCT05362409
Title: A Phase 1 Multi-center Clinical Trial Evaluating the Safety and Tolerability of 5-aminolevulinic Acid (5-ALA) Combined With CV01 Delivery of Ultrasound for Sonodynamic Therapy(SDT) in Patients With Recurrent High Grade Glioma (HGG)
Brief Title: Study to Evaluate 5-ALA Combined With CV01 Delivery of Ultrasound in Recurrent High Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alpheus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CV01-101
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-01

CONDITIONS: High Grade Glioma
Keywords: Cancer; Brain Cancer; Sonodynamic; Glioma; High Grade Glioma (HGG); Sonodynamic therapy (SDT); Glioblastoma
MeSH Terms: conditions — Glioma; Neoplasms; Brain Neoplasms; Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: Part A will include cohorts at escalating duration of sonication. Parts B and C will include the recommended duration as determined in Part A.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- 5-ALA with CV01 (Experimental): 5-aminolevulinic acid [5-ALA] with CV01-delivered ultrasound
  Interventions: Drug: 5 Aminolevulinic Acid; Device: CV01-delivered ultrasound

INTERVENTIONS:
Drug: 5 Aminolevulinic Acid — 5-aminolevulinic acid [5-ALA] administered orally 20 mg/kg every 4 weeks
  Other Names: 5-ALA; Gleolan
Device: CV01-delivered ultrasound — CV01-delivered ultrasound every 4 weeks

SUMMARY:
A Phase 1 Multi-center clinical Trial Evaluating the Safety and Tolerability of 5-aminolevulinic Acid (5-ALA) Combined With CV01 Delivery of Ultrasound for Sonodynamic Therapy (SDT) in Patients With recurrent High Grade Glioma (HGG).

DETAILED DESCRIPTION:
High-grade gliomas are the most commonly occurring primary CNS tumors in adults. The investigational product in this clinical study is a drug-device combination product consisting of 5-ALA HCl oral solution and the CV01 ultrasound delivery device. 5-ALA will be administered as a sonosensitizer prior to CV01-delivered ultrasound and will be re-administered every 4 weeks prior to CV01 ultrasound delivery. The CV01 device will deliver non-ablative, low-intensity ultrasound to deep regions of the brain to induce apoptosis of cancer cells. Part A will focus on duration escalation and determining the recommended duration of CV01 delivered ultrasound. Part B will further explore safety and tolerability through cohort expansion at the recommended duration of CV01 delivered ultrasound. Part C will include an exploratory surgical cohort at the recommended duration of CV01 delivered ultrasound. This FIH study will evaluate escalating durations of ultrasound delivery with CV01 and will enroll up to 48 patients.

ELIGIBILITY:
Key Inclusion Criteria

1. Patient must provide informed consent, stating understanding of the procedures and investigational nature of the study treatment, and willingness to comply with study requirements
2. ≥ 18 years of age
3. WHO performance status of ≤ 2 at screening
4. Part A: Previous histopathologically confirmed diagnosis of high-grade glioma and radiographic evidence of recurrence after prior therapy with radiotherapy. Eligible histologies include (according to WHO classification 2021):

   1. Astrocytoma, WHO grade 3 and 4 (including subtypes)
   2. Oligodendroglioma WHO grade 3 (including subtypes)

   Parts B and C: Previous histopathologically confirmed diagnosis of glioblastoma and radiographic evidence of recurrence after prior therapy with radiotherapy. While Part A may include patients with any type of HGG and any number of recurrences, Parts B and C are restricted to patients with glioblastoma experiencing first recurrence.
5. Unifocal or multifocal tumor confined to the supratentorial compartment
6. Interval since last anti-cancer therapy relative to first 5-ALA treatment, as detailed below

   1. End of radiotherapy >12 weeks (including skin-directed radiation for skin cancer),
   2. Last cytotoxic chemotherapy (4 weeks, if prior nitrosureas 6 weeks).
   3. Last biological therapy, i. If bevacizumab ≥ 6 weeks ii. If other monoclonal antibody, e.g., immune checkpoint inhibitor > 3 weeks iii. If tyrosine kinase inhibitor or other small molecule > 2 weeks
   4. Any other investigational agent(s) ≥ 30 days or 5 half-lives, whichever is longer
   5. Photodynamic therapy for skin cancer or actinic keratoses ≥ 12 weeks
7. Any toxicity attributable to prior anti-cancer therapy must be resolved to the patient's baseline level or ≤ Grade 1 (except alopecia).
8. Adequate bone marrow and organ function, defined by the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥ 1000 cells/mm3
   2. Platelet count ≥ 100,000 cells/mm3
   3. Hemoglobin (Hgb) ≥ 8 g/dL
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
   5. Total bilirubin ≤ 1.5 x ULN (unless Gilbert's syndrome, then patients may be eligible if total serum bilirubin is ≤ 3.0 x ULN or direct bilirubin is ≤ 1.5 x ULN)
   6. Creatinine clearance (CrCL) as estimated by Cockcroft-Gault equation of ≥ 50 mL/min
9. Adequate coagulation function defined as PT (prothrombin time)/PTT (partial thromboplastin time) within normal institutional values
10. Males or non-pregnant, non-lactating females who are postmenopausal, surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation or hysterectomy), or who agree to use effective contraceptive methods as defined by the protocol during the study and for 30 days after the last investigational treatment, see Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea and a serum follicle stimulating hormone (FSH) concentration ≥ 40 IU/L, or at least 6 weeks following surgical menopause (bilateral oophorectomy).

    a. Women of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) pregnancy test within 7 days prior to first 5-ALA administration
11. Agreement to adhere to Lifestyle Considerations throughout study duration
12. Part C, Surgical group only: Tumor resection surgery is clinically indicated and planned for the patient, regardless of study participation

Key Exclusion Criteria:

1. Primary infratentorial or brainstem tumors
2. Primary spinal cord tumors
3. Bihemispheric disease (enhancing or non-enhancing) or tumors that involve the bilateral corpus callosum
4. Women who are pregnant or breastfeeding
5. Inability to undergo MRI or receive gadolinium (Gd)-based contrast agents
6. Hypersensitivity to 5-ALA or porphyrins
7. Average skull thickness at the treatment field > 10 mm as assessed by Alpheus Medical.

   The treatment field is defined as the various locations on the head where the transducer will be coupled to the patient. The average skull thickness at each treatment field will be determined by Alpheus Medical through post-processing the thin cut head computed tomography (CT) (without contrast). The patient's CT scan must be provided to Alpheus Medical for evaluation as part of the Screening and Enrollment process.
8. Hemorrhagic or ischemic stroke (including transient ischemic attacks) and central nervous system bleeding in the preceding 6 months that are not related to glioma surgery. History of prior intratumoral bleeding is not an exclusion criterion; however, patients with a history of prior intratumoral or intracranial bleeding will undergo a non-contrast head CT to exclude acute bleeding.
9. Patients who have clinically significant edema requiring urgent intervention (e.g., surgery, initiation of steroids, escalating doses of steroids).
10. Patients with progressive and rapid clinical deterioration that, in the opinion of the investigator, is likely to worsen during the first cycle of treatment or in the peri-operative interval (in the surgical cohort)
11. Cumulative prior RT dose > 64 Gy
12. Acute or chronic types of porphyria
13. Gastrointestinal disorder that negatively affects absorption
14. Known active hepatitis B or C (Note: testing is not required)
15. Known human immunodeficiency virus (HIV) infection (Note: testing is not required)
16. Unable to avoid phototoxic drugs (e.g., St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulfonamides, quinolones, and tetracyclines) for 24 hours prior to and following 5-ALA administration
17. Any other concurrent severe or uncontrolled concomitant medical condition that could compromise participation in the study (e.g., clinically significant pulmonary disease, cardiac disease, clinically significant psychiatric or neurological disorder, active or uncontrolled infection)
18. Patient has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (Safety and Tolerability) | 12 Months
  Safety and tolerability as determined by the incidence of adverse events (AEs), including severe AEs and serious AEs (SAEs)
To determine the Maximum Tolerable Duration (MTDu) | 12 Months
  The MTDu is defined as the highest duration at which fewer than 1/3 of patients experience a Duration limited toxicity

SECONDARY OUTCOMES:
Assessment of Overall response rate (ORR) | 12 Months
  ORR assessed by RANO criteria
Assessment of Duration of Response (DoR) | 12 Months
Assessment of Overall survival (OS) | 12 Months
Assessment of Progression free survival (PFS) | 12 Months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Washington University School of Medicine in St.Louis, St Louis, Missouri
  - Dent Neurosciences Research Center, Amherst, New York
  - Northwell, Lake Success, New York

IPD SHARING:
Plan to Share IPD: No